CLINICAL TRIAL: NCT00000660
Title: Phase I Study of Weekly Oral VP-16 for AIDS-Associated Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 110; 11085 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Drug Evaluation; Etoposide; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Etoposide

INTERVENTIONS:
Drug: Etoposide

SUMMARY:
To define the toxicity and maximum-tolerated dose of weekly oral etoposide (VP-16) in patients with AIDS-related Kaposi's sarcoma; to determine the clinical pharmacology of orally administered VP-16 in AIDS patients. A secondary objective is to obtain preliminary data for determining the effect of oral VP-16 on Kaposi's sarcoma.

VP-16 is an antitumor agent. Previous problems with VP-16 include the route of administration and the toxicities. VP-16 has been given intravenously for 3 consecutive days in a 21-day cycle for lung cancer and testicular cancer. VP-16 has also been used in lymphoma therapy. Oral VP-16 would eliminate the need for an intravenous catheter and so a patient could avoid the pain, inconvenience, and potential complications associated with medications administered intravenously. The relative ease of outpatient administration and the potentially significant antitumor activity of oral VP-16 motivates this study. The possibility of weekly drug administration is the other focus of this study.

DETAILED DESCRIPTION:
VP-16 is an antitumor agent. Previous problems with VP-16 include the route of administration and the toxicities. VP-16 has been given intravenously for 3 consecutive days in a 21-day cycle for lung cancer and testicular cancer. VP-16 has also been used in lymphoma therapy. Oral VP-16 would eliminate the need for an intravenous catheter and so a patient could avoid the pain, inconvenience, and potential complications associated with medications administered intravenously. The relative ease of outpatient administration and the potentially significant antitumor activity of oral VP-16 motivates this study. The possibility of weekly drug administration is the other focus of this study.

Four patients are entered at each dose level starting with level 1. Patients are not entered into the next higher dose level until at least two patients at the previous dose level have completed at least 3 weeks of therapy with grade 2 or less maximum tolerated dose-defining toxicities. Treatment is repeated weekly for 52 weeks until either a grade 3 or 4 toxicity occurs, or until a patient shows a complete response or progressive disease. Patients with a complete response are continued on drug for 4 additional weeks from the time that complete response is first documented. Patients with progressive disease are withdrawn from study. Patients with partial response or stable disease continue until either unacceptable toxicity occurs or a complete response or progression of disease is reached.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

AMENDED:

* 04-21-91 Zidovudine (AZT) allowed after completing 8 weeks on the study. Patients on reduced doses of VP-16 must have tolerated at least 4 consecutive weeks at the reduced dose before starting AZT. Zidovudine will not be provided by the NIAID Clinical Product Research Repository.

AMENDED:

* Zidovudine (AZT) allowed after completing 12 weeks on study.

Allowed:

* Aerosolized pentamidine for Pneumocystis carinii pneumonia prophylaxis (PCP).

Concurrent Treatment:

Allowed:

* Local radiotherapy or laser therapy to cosmetically apparent, non-indicator lesions provided the dose to any one lesion does not exceed 300 rads and the total surface area of all lesions treated does not exceed 10 cm2.

Risk Behavior:

Allowed:

* All risk groups.

Patients must:

* Have AIDS-related Kaposi's sarcoma.
* Be ineligible for protocols of higher priority at study center.
* Be willing to sign an informed consent or have guardian willing to sign.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active opportunistic infection not specifically allowed.
* Concurrent neoplasm not specifically allowed.
* Significant neurologic, cardiac, or liver disease.

Concurrent Medication:

Excluded:

* Therapy with potentially myelosuppressive, hepatotoxic, or nephrotoxic drugs for an opportunistic infection.

Patients with the following are excluded:

* Active opportunistic infection not specifically allowed.
* Ongoing therapy, including maintenance therapy, for an opportunistic infection with potentially myelosuppressive, hepatotoxic, or nephrotoxic drugs.
* Concurrent neoplasm not specifically allowed.
* Significant neurologic, cardiac, or liver disease.

Prior Medication:

Excluded:

* Biologic response modifiers or corticosteroids within 14 days prior to study entry.
* Cytotoxic chemotherapy within 30 days prior to study entry.
* Ribavirin within 6 weeks prior to study entry.
* Azidothymidine (AZT), alpha-interferon, didanosine (ddI), ganciclovir (DHPG), or any other antiretroviral drugs within 1 week prior to study entry.

Prior Treatment:

Excluded within 30 days prior to study entry:

* Radiation therapy with > 4000 rads.
* Total skin electron beam therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 1992-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Kahn, Study Chair; S Krown, Study Chair
Locations (6):
- United States (6):
  - San Francisco Gen Hosp, San Francisco, California
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Paredes J, Kahn JO, Tong WP, Feldstein ML, Lin S, Bennett JM, Metroka CE, Ratner L, Krown SE. Weekly oral etoposide in patients with Kaposi's sarcoma associated with human immunodeficiency virus infection: a phase I multicenter trial of the AIDS Clinical Trials Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Jun 1;9(2):138-44. PMID 7749790